CLINICAL TRIAL: NCT01773889
Title: A Phase II Trial of Intravenous Denileukin Diftitox Plus Subcutaneous Pegylated IFNα-2a to Treat Epithelial Ovarian Cancer FIGO Stage III or Stage IV, Extraovarian Peritoneal or Fallopian Tube Carcinoma or Ineligible for First-Line Therapy
Brief Title: A Trial of Intravenous Denileukin Diftitox Plus Subcutaneous Pegylated IFNα-2A in Stage III or IV Ovarian Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC20090233H; OCR 09-01 (Other: UTHSCSA)
Record Dates: First submitted 2013-01-14; First posted 2013-01-23 (Estimated); Results first posted 2013-07-02 (Estimated); Last update posted 2018-04-10 (Actual); Status verified 2013-05

CONDITIONS: Epithelial Ovarian Cancer; Extraovarian Peritoneal Cancer; Fallopian Tube Carcinoma
Keywords: Epithelial Ovarian Cancer; FIGO (Int Federation of Gyn and Ob )Stage III or Stage IV; Extraovarian Peritoneal Cancer; Fallopian Tube Carcinoma Failing
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Fallopian Tube Neoplasms | interventions — denileukin diftitox

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Denileukin Diftitox/SC Pegylated IFNα-2A (Experimental): Administration of Denileukin Diftitox Plus Subcutaneous Pegylated IFNα-2A
  Interventions: Drug: Denileukin Diftitox/SC Pegylated IFNα-2a

INTERVENTIONS:
Drug: Denileukin Diftitox/SC Pegylated IFNα-2a
  Other Names: Ontak plus Pegylated IFNα-2a

SUMMARY:
This study will test the hypothesis that adding pegylated IFN (IFN)a-2b to denileukin diftitox improves the potential of denileukin diftitox alone to deplete regulatory T cells (Tregs) and will thereby boost tumor immunity in patients with advanced-stage epithelial ovarian cancers, enhancing treatment efficacy.

DETAILED DESCRIPTION:
The aims of this study are to:

* Assess the efficacy of adding pegylated IFN-α2b to denileukin diftitox to treat selected advanced-stage epithelial ovarian cancers
* Test the immune-modulating effects of adding pegylated IFN-α2b to denileukin diftitox in ovarian cancer patients and relate them to clinical efficacy
* Identify any toxicity associated with pegylated IFN-α2b plus denileukin diftitox treatment in these patients
* Identify practical means to dose the immunomodulating agents denileukin diftitox and pegylated IFN-α2b based on immunopharmacodynamic metrics

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent
* Not on immune-modulating drugs, except those used as denileukin diftitox premedication, unless the principal investigator grants an exception (which exception must be documented in writing)
* Histologically proven epithelial (non-germ cell, non-stromal cell) cancer of the ovaries, fallopian tubes or extraovarian peritoneal carcinoma. Clinical recurrence without documented pathology is acceptable
* FIGO stage III or IV with failed prior first-line therapy, or ineligible for or intolerant of such therapy
* Measurable disease as defined in section 6 within 30 days of study enrollment
* Blood hemoglobin ≥ 8.5 gm/dl within 7 days of study enrollment
* Absolute neutrophil count ≥ 750/mm3 within 7 days of study enrollment
* Platelet count ≥ 40,000/mm3 within 7 days of study enrollment
* SGOT (serum glutamic oxaloacetic transaminase) ≤10 x upper limit of normal within 7 days of study enrollment
* Normal TSH (thyroid-stimulating hormone ) within 30 days of study enrollment
* No chemotherapy in the 14 days prior or radiation therapy in the thirty days prior to initiation of treatment on this study
* No other concurrent chemotherapy, surgery or radiation therapy during this protocol except surgery or radiation therapy to control symptoms with concurrence of the principal investigator
* No contraindication to any study treatment
* No active major medical problems, including untreated or uncontrolled infections
* Beck Depression Index ≥15 within 30 days of study enrollment
* If of reproductive potential, a negative urine pregnancy test within 3 days of study enrollment, and agreement to use adequate contraception. Pregnancy testing will continue monthly while on treatment unless the subject is no longer able to become pregnant or there is sufficient justification otherwise
* Not breast feeding
* Life expectancy ≥ six months
* ECOG (Eastern Cooperative Oncology Group) performance status ≤ 2
* Serum albumin ≥ 1.8 gm/dl
* Age ≥ 18 years
* Acceptable baseline retinal examination within 30 days of study enrollment
* No active substance abuse in the prior 6 months
* Patients failing single agent denileukin diftitox in the ongoing trial "A Phase II Trial of Intravenous Ontak to Treat Epithelial Ovarian Cancer FIGO Stage III or Stage IV, or Extraovarian Peritoneal Carcinoma, Failing or Ineligible for First-Line Therapy" are eligible for this trial provided that three or more weeks have elapsed since their last denileukin diftitox infusion and they meet all eligibility criteria and successfully undergo all screening examinations for this trial.

Exclusion Criteria:

* Unable to tolerate phlebotomy
* Germ cell or stromal cell cancers of the ovaries, or other currently uncured cancer
* Active autoimmune disease including systemic lupus erythematosus, psoriasis, or inflammatory bowel disease that is not medically controlled
* Autoimmune hepatitis, whether medically controlled or not
* Contraindication to any study drug
* Known hypersensitivity to denileukin diftitox, pegylated IFN-α2a or any of their components or excipients
* Current pregnancy or breast feeding
* Inability to document adequate contraception if a female of reproductive potential
* On other immune-modulating drugs, except denileukin diftitox premedications or those approved by the principal investigator
* Chemotherapy within 14 days or radiation therapy within the thirty days prior to initiation of study treatment
* Life expectancy less than six months
* Serum albumin < 1.8 gm/dl
* Blood hemoglobin < 8.5 gm/dl
* ECOG performance status> 2
* Symptomatic coronary artery disease (including uncontrolled angina, congestive heart failure, and the like)
* Uncontrolled hypertension (diastolic BP consistently >100 mm Hg or systolic BP consistently >160 mm Hg on a regular basis)
* Uncontrolled, symptomatic cardiac arrhythmia
* Retinopathy associated with significant visual impairment
* Beck Depression Index >15
* Active substance abuse in the prior 6 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2009-06; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tyler Curiel, MD, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- CTRC (Cancer Therapy and Research Center) at UTHSCSA, San Antonio, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was open to accrual on 7/29/2009 and closed to accrual on 6/27/2011. Subjects were seen at The Cancer Therapy and Research Center @ The University of Texas Health Science Center San Antonio.
Pre-assignment Details: * Intercurrent illness that prevents further administration of treatment
  * Unacceptable adverse event(s)
  * Patient withdraws from study
  * General or specific changes in the patient's condition render the patient unacceptable for further treatment in the judgment of the investigator.
Groups:
- Denileukin Diftitox Plus Subcutaneous Pegylated IFNα-2A: Denileukin Diftitox Plus Subcutaneous Pegylated IFNα-2a :
Period: Overall Study
Arm/Group | Denileukin Diftitox Plus Subcutaneous Pegylated IFNα-2A
Started | 2
Completed | 0
Not Completed | 2
Not completed — lack of funding | 2

BASELINE CHARACTERISTICS:
Arm/Group | Denileukin Diftitox Plus Subcutaneous Pegylated IFNα-2A
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Clinical Response Rate
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Response = CR + PR.
  Failure to respond criteria are not based on RECIST criteria, which have unclear application to immune-based clinical trials. Instead, novel lack-of-failure criteria, rather than failure-of-success criteria have been written to avoid stopping therapy prematurely without compromising patient safety, to accommodate the uncertainties of assessing failure in this setting. The criteria as written are based on sound medical, scientific and ethical principles. The trial is further designed to help establish the utility of these novel criteria.
Time Frame: every 3 months until the date of first documented progression or date of death from any cause, assessed up to 2 years when study terminated early
Measure: Number; unit: participants
Arm/Group | Denileukin Diftitox Plus Subcutaneous Pegylated IFNα-2A
Number analyzed (Participants) | 2
participants | 2

ADVERSE EVENTS:
Arm/Group | Denileukin Diftitox Plus Subcutaneous Pegylated IFNα-2A
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No